CLINICAL TRIAL: NCT01230983
Title: Intensive Treatment For T-CELL Acute Lymphoblastic Leukemia and Advanced Stage Lymphoblastic Non-Hodgkin's Lymphoma: A Pediatric Oncology Group Phase III Study
Brief Title: Combination Chemotherapy in Treating Patients With Acute Lymphoblastic Leukemia or Advanced Lymphoblastic Non-Hodgkin's Lymphoma
Acronym: T-Cell #4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 9404; U10CA030969 (NIH); POG-9404 (Other: Pediatric Oncology Group); CDR0000064664 (Other: Clinical Trials.gov)
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Cardiac Toxicity; Leukemia; Lymphoma
Keywords: stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; untreated childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; cardiac toxicity
MeSH Terms: conditions — Cardiotoxicity; Leukemia; Lymphoma | interventions — Asparaginase; Cytarabine; Dexrazoxane; Razoxane; Doxorubicin; Leucovorin; Mercaptopurine; Methotrexate; Prednisone; Hydrocortisone; hydrocortisone hemisuccinate; Vincristine; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment 1: (No HD MTX / No Zinecard) (Experimental): Closed 09/2000 Induction (Vincristine sulfate, Prednisone, doxorubicin hydrochloride, Methotrexate (MTX), mercaptopurine (6-MP), methotrexate/cytarabine), Consolidation (Vincristine sulfate), Prednisone, doxorubicin hydrochloride, mercaptopurine (6-MP), asparaginase, IT methotrexate /cytarabine radiation therapy (XRT)). Continuation (Vincristine sulfate, Prednisone, IT methotrexate/Ara-C,mercaptopurine (6-MP), IT methotrexate/cytarabine)
  Interventions: Drug: asparaginase; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: radiation therapy
- Treatment 2: (No HD MTX / Zinecard) (Active Comparator): Closed 09/2000 Induction (Vincristine sulfate, Prednisone, doxorubicin hydrochloride, Methotrexate (MTX), mercaptopurine (6-MP), methotrexate/cytarabine, dexrazoxane hydrochloride (Zinecard or DZR)), Consolidation (Vincristine sulfate), Prednisone, doxorubicin hydrochloride, mercaptopurine (6-MP), asparaginase, dexrazoxane hydrochloride (Zinecard or DZR), IT methotrexate /cytarabine, radiation therapy (XRT)). Continuation (Vincristine sulfate, Prednisone, IT methotrexate/Ara-C,mercaptopurine (6-MP), IT methotrexate/cytarabine)
  Interventions: Drug: asparaginase; Drug: cytarabine; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: radiation therapy
- Treatment 3: (HD MTX / No Zinecard) (Active Comparator): Closed 09/2001 Induction (Vincristine sulfate, Prednisone, doxorubicin hydrochloride, Methotrexate (MTX), mercaptopurine (6-MP), leucovorin calcium (LCV), HD methotrexate/cytarabine), Consolidation (Vincristine sulfate), Prednisone, doxorubicin hydrochloride, mercaptopurine (6-MP), asparaginase, leucovorin calcium (LCV), HD methotrexate /cytarabine radiation therapy (XRT)). Continuation (Vincristine sulfate, Prednisone, IT methotrexate/Ara-C,mercaptopurine (6-MP), HD methotrexate/cytarabine)
  Interventions: Drug: asparaginase; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: radiation therapy
- Treatment 4: (HD MTX / Zinecard) (Active Comparator): Closed 09/2001 Induction (Vincristine sulfate, Prednisone, doxorubicin hydrochloride, Methotrexate (MTX), mercaptopurine (6-MP), leucovorin calcium (LCV), HD methotrexate/cytarabine, dexrazoxane hydrochloride (Zinecard or DZR)), Consolidation (Vincristine sulfate), Prednisone, doxorubicin hydrochloride, mercaptopurine (6-MP), asparaginase, HD methotrexate /cytarabine, dexrazoxane hydrochloride (Zinecard or DZR), radiation therapy (XRT)). Continuation (Vincristine sulfate, Prednisone, IT methotrexate/Ara-C,mercaptopurine (6-MP), HD methotrexate/cytarabine)
  Interventions: Drug: asparaginase; Drug: cytarabine; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: asparaginase — Given IV
  Other Names: E. coli; Elspar; NSC #10922
Drug: cytarabine — Given IV
  Other Names: Cytosine Arabinoside; AraC; Cytosar; NSC #06387
Drug: dexrazoxane hydrochloride — Given IV
  Other Names: DZR; ADR-529; ZINECARD; ICRF-187; NSC #169780
  Arms: Treatment 2: (No HD MTX / Zinecard); Treatment 4: (HD MTX / Zinecard)
Drug: doxorubicin hydrochloride — Given IV
  Other Names: Doxorubicin; NSC #123127
Drug: leucovorin calcium — Given IV
  Other Names: LCV; Wellcovorin; citrovorum factor; folinic acid; NSC #003590
  Arms: Treatment 3: (HD MTX / No Zinecard); Treatment 4: (HD MTX / Zinecard)
Drug: mercaptopurine — Given orally
  Other Names: 6-MP; Purinethol; NSC #000755
Drug: methotrexate — Given IV
  Other Names: MTX; amethopterin; NSC #000740
Drug: prednisone — Given orally
  Other Names: Deltasone; Meticorten; Liquid Pred; NSC #010023
Drug: therapeutic hydrocortisone — Given IT
  Other Names: hydrocortisone sodium succinate; Solu-cortef; NSC #010483
Drug: vincristine sulfate — Given IV
  Other Names: VCR; Oncovin; NSC #067574
Radiation: radiation therapy — Radiation to cranium
  Other Names: XRT

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Dexrazoxane may lessen the side effects of chemotherapy.

PURPOSE: Randomized phase III trial to compare combination chemotherapy with or without dexrazoxane and with or without high-dose methotrexate in patients with acute lymphoblastic leukemia or advanced lymphoblastic non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine, in a randomized trial, the effectiveness of high-dose methotrexate when added to a multiagent chemotherapy backbone (the Dana Farber Cancer Institute regimen, protocol DFCI-87001) proven effective in T-cell acute lymphoblastic leukemia (T-ALL) and advanced lymphoblastic non-Hodgkin's lymphoma (NHL). II. Determine the role of dexrazoxane in preventing cardiotoxicity in children with T-ALL and advanced lymphoblastic NHL treated with an anthracycline-based regimen. III. Study the biology of T-cell lymphoid malignancies by accumulating data on the concurrent ALL classification study (POG-9400) and analyzing the data relative to outcome. IV. Evaluate the correlation of minimal residual disease (using the TAL 1 proto-oncogene) with event-free survival. V. Determine the role of p53 and p16 tumor suppressor genes in T-ALL. VI. Determine whether drug sensitivity profiles of blast cells to doxorubicin, methotrexate, and cytarabine correlate with initial response and subsequent relapse.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease category (acute lymphoblastic leukemia (ALL) with no CNS disease vs. ALL with CNS disease vs. non-Hodgkin's lymphoma (NHL) with no CNS disease vs. NHL with CNS disease), gender, race (Caucasian vs. African American vs. Hispanic). Patients are randomized to one of four treatment arms. ARM I: During induction therapy, patients receive vincristine IV once daily on days 1, 8, 15, and 22, oral prednisone three times a day on days 1-21, doxorubicin IV daily on days 1, 2, and 22, methotrexate IV once, at least 8 hours after doxorubicin on day 2, and oral mercaptopurine daily on days 22-35. Patients receive triple intrathecal therapy (TIT) consisting of methotrexate, cytarabine, and hydrocortisone on weeks 1, 3, 4, 5, and 6. Patients with CNS 2 or 3 disease receive TIT on week 2. During weeks 7-33, patients receive consolidation therapy consisting of vincristine IV once every 3 weeks, oral prednisone three times a day over 5 days, every 3 weeks, doxorubicin IV once every 3 weeks, oral mercaptopurine daily for 14 days, every 3 weeks, and asparaginase intramuscularly (IM) weekly on weeks 7-26. Patients receive TIT on week 10 and 22 (on week 16 for patients with CNS 2 or 3 disease). Patients receive radiotherapy beginning on week 22. During weeks 34-108, patients receive continuation therapy consisting of vincristine IV once every 3 weeks, oral prednisone three times a day over 5 days, every 3 weeks, methotrexate IV or IM weekly (omitted during TIT) and oral mercaptopurine daily for 14 days, every 3 weeks. Patients receive TIT on weeks 40, 58, 76, and 94. Arm II: Patients receive induction therapy as in Arm I with an addition of dexrazoxane IV given prior to doxorubicin on days 1, 2, and 22. Patients receive consolidation therapy as in Arm I with an addition of dexrazoxane IV given prior to doxorubicin once every 3 weeks. Patients receive continuation therapy as in Arm I. Arm III: Patients receive induction therapy as in Arm I in addition to high dose methotrexate IV on week 4 and leucovorin calcium IV or orally every 6 hours for 7 doses beginning 36 hours after high dose methotrexate. Patients receive consolidation therapy as in Arm I in addition to high dose methotrexate IV on weeks 7, 10, and 13 followed by leucovorin calcium as in induction therapy. Patients receive continuation therapy as in Arm I. Arm IV: Patients receive induction therapy and consolidation therapy as in Arms I, II, and III. Patients receive continuation therapy as in Arm I. Treatment continues for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 2 months for 1 year, every 4 months for 3 years, then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 494 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: T-cell acute lymphoblastic leukemia (ALL) Registration on current ALL classification study (POG-9400) required within 6 working days prior to entry DR-, T+ DR-, T- or DR+, T+ eligible if T-cell ALL confirmed at the Johns Hopkins Reference Laboratory Biopsy-proven diffuse lymphoblastic lymphoma Murphy stage III/IV disease Registered on ALL classification study (POG-9400)

PATIENT CHARACTERISTICS: Age: Over 12 months to under 22 years for T-ALL Under 22 years for lymphoma

PRIOR CONCURRENT THERAPY: No prior therapy other than steroids or emergency mediastinal irradiation in patients with severe respiratory distress from mediastinal disease Steroid treatment allowed provided that physical examination and complete blood count with differential were performed immediately prior to beginning steroids and results of both are known

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 573 (Actual)
Dates: Start 1996-06; Primary Completion 2001-09 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Complete Continuous Remission | Time to failure for any cause among patients achieving a complete response
  Since all patients receive the same induction, the endpoint will be CCR , i.e. complete continuous remission (the time to failure for any cause among patients achieving a complete response)

SECONDARY OUTCOMES:
Abnormalities in the 31 week and the year 3 echocardiograms | 1 year off therapy
  Endpoint will be abnormalities in the 31 week and the year 3 echocardiograms (i.e. year 1 off therapy). Secondarily, we shall compare the CCR rates for the two treatment regimens, in a two sided fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L. Asselin, MD, Study Chair — James P. Wilmot Cancer Center

REFERENCES:
- [Background] Cleaver AL, Beesley AH, Firth MJ, Sturges NC, O'Leary RA, Hunger SP, Baker DL, Kees UR. Gene-based outcome prediction in multiple cohorts of pediatric T-cell acute lymphoblastic leukemia: a Children's Oncology Group study. Mol Cancer. 2010 May 12;9:105. doi: 10.1186/1476-4598-9-105. PMID 20459861
- [Background] Salzer WL, Devidas M, Carroll WL, Winick N, Pullen J, Hunger SP, Camitta BA. Long-term results of the pediatric oncology group studies for childhood acute lymphoblastic leukemia 1984-2001: a report from the children's oncology group. Leukemia. 2010 Feb;24(2):355-70. doi: 10.1038/leu.2009.261. Epub 2009 Dec 17. PMID 20016527
- [Background] Matloub Y, Asselin BL, Stork LC, et al.: Outcome of children with T-Cell acute lymphoblastic leukemia (T-ALL) and standard risk (SR) features: results of CCG-1952, CCG-1991 and POG 9404. [Abstract] Blood 104 (11): A-680, 195a, 2004.
- [Background] Seibel NL, Asselin BL, Nachman JB, et al.: Treatment of high risk T-cell acute lymphoblastic leukemia (T-ALL): comparison of recent experience of the Children's Cancer Group (CCG) and Pediatric Oncology Group (POG). [Abstract] Blood 104 (11): A-681, 2004.